CLINICAL TRIAL: NCT07396311
Title: Fractional Exhaled Nitric Oxide (FeNO) as a Predictor of Exacerbations in COPD Patients Initiated on Triple Inhaler Therapy: A Prospective Exploratory Cohort Study
Brief Title: Fractional Exhaled Nitric Oxide and Exacerbations of COPD
Status: Not yet recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2512090251
Record Dates: First submitted 2026-02-01; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; FeNO; Triple Inhaler Therapy; Exacerbation; Air Pollution; Type 2 Inflammation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD Patients Initiated on Triple Inhaler Therapy: This cohort includes patients with chronic obstructive pulmonary disease (COPD) receiving triple inhaler therapy (inhaled corticosteroid/long-acting beta-agonist/long-acting muscarinic antagonist) as part of routine clinical care following one or more recent exacerbations. Eligible participants include both patients who have been escalated to triple therapy due to prior exacerbations and are already receiving triple therapy at enrollment, as well as patients who are newly prescribed triple therapy at or immediately before enrollment because of a recent exacerbation. All participants are followed prospectively for up to 12 months to assess exacerbations, lung function, symptoms, and inflammatory biomarkers. Baseline fractional exhaled nitric oxide (FeNO) is evaluated as a predictor of clinical outcomes.
  Interventions: Other: No intervention assigned

INTERVENTIONS:
Other: No intervention assigned — No investigational intervention is assigned in this observational study. All treatments, including triple inhaler therapy, are prescribed at the discretion of the treating physicians as part of routine clinical care. The research team does not assign, modify, or mandate any therapeutic intervention.

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a heterogeneous condition with recurrent exacerbations despite guideline-based therapy. This prospective observational cohort study aims to evaluate whether baseline fractional exhaled nitric oxide (FeNO), a biomarker of type 2 airway inflammation, predicts future exacerbations and lung function decline in COPD patients initiated on triple inhaler therapy in routine clinical practice. The study will also explore the relationships between air pollution exposure, type 2 inflammatory biomarkers, and COPD outcomes.

DETAILED DESCRIPTION:
This is a pragmatic, prospective, longitudinal observational cohort study conducted in patients with COPD who are initiated on triple inhaler therapy as part of routine clinical care. No investigational drugs, devices, or protocol-mandated interventions are administered. Biomarker measurements, including fractional exhaled nitric oxide (FeNO), are performed for research purposes only and do not influence clinical decision-making.

Participants will be followed for up to 12 months after enrollment with scheduled assessments of exacerbation events, lung function, symptom burden, and biomarkers. The total study duration is approximately 24 months, accounting for a 12-month enrollment period and completion of follow-up for the last enrolled participant. Environmental air pollution exposure will be estimated using a validated hybrid kriging/land-use regression model based on residential address.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 40 years or older
* Diagnosis of chronic obstructive pulmonary disease (COPD) confirmed by post-bronchodilator spirometry (FEV₁/FVC < 0.70).
* History of cigarette smoking
* Receiving triple inhaler therapy (inhaled corticosteroid/long-acting beta-agonist/long-acting muscarinic antagonist) as part of routine clinical care, including:
* patients who have been previously escalated to triple inhaler therapy due to prior exacerbations and are already receiving triple therapy at the time of enrollment, and
* patients who are newly prescribed triple inhaler therapy at or immediately before enrollment because of a recent exacerbation.

Exclusion Criteria:

-

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are recruited from adult COPD patients receiving routine pulmonary care at a tertiary hospital outpatient clinic, including follow-up visits after exacerbations and referrals from primary or emergency care.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-02-29 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Annualized rate of moderate-to-severe COPD exacerbations | Up to 12 months after enrollment
  Moderate exacerbations are defined as those requiring systemic corticosteroids, antibiotics, or both. Severe exacerbations are defined as those requiring hospitalization or emergency department visits lasting more than 24 hours.

SECONDARY OUTCOMES:
Change in lung function (FEV₁) | Up to 12 months after enrollment
  Rate of decline in pre-bronchodilator FEV₁
Change in COPD Assessment Test (CAT) score | Up to 12 months after enrollment
  Change in symptom burden assessed by CAT

OTHER OUTCOMES:
Multimarker and Environmental Interaction | up to 12 months
  Multivariable negative binomial models will include FeNO (spline + categories), eosinophils (<100, 100-<300, ≥300 cells/µL), IgE (log-transformed), and air pollutants (PM10, PM2.5, NO2, SO2, CO, and O3; levels of baseline, 1-month, 6-month, and 1-year follow-up). FeNO-specific adjusted IRRs and predicted rates at 15, 20, 25, 35, and 50 ppb will be presented. Significant interactions (FeNO×smoking, FeNO×ICS dose, FeNO×PM₂.₅ quartiles) will be visualized with stratum-specific curves.
  This analysis will determine whether FeNO remains a consistent predictor across different inflammatory or environmental contexts, or whether its predictive value varies depending on eosinophil counts, smoking status, or air pollution exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Ting-Yu Lin, MD., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Medical Foundation, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. The study involves clinical and environmental data that may pose a risk of re-identification despite de-identification, and no data-sharing infrastructure is currently established.

REFERENCES:
- [Background] Papi A, Romagnoli M, Baraldo S, Braccioni F, Guzzinati I, Saetta M, Ciaccia A, Fabbri LM. Partial reversibility of airflow limitation and increased exhaled NO and sputum eosinophilia in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2000 Nov;162(5):1773-7. doi: 10.1164/ajrccm.162.5.9910112. PMID 11069811
- [Background] Alcazar-Navarrete B, Ruiz Rodriguez O, Conde Baena P, Romero Palacios PJ, Agusti A. Persistently elevated exhaled nitric oxide fraction is associated with increased risk of exacerbation in COPD. Eur Respir J. 2018 Jan 18;51(1):1701457. doi: 10.1183/13993003.01457-2017. Print 2018 Jan. PMID 29348180
- [Background] Zhou A, Zhou Z, Deng D, Zhao Y, Duan J, Cheng W, Liu C, Chen P. The Value of FENO Measurement for Predicting Treatment Response in Patients with Acute Exacerbation of Chronic Obstructive Pulmonary Disease. Int J Chron Obstruct Pulmon Dis. 2020 Sep 24;15:2257-2266. doi: 10.2147/COPD.S263673. eCollection 2020. PMID 33061343
- [Background] Romero-Linares A, Alvarez-Muro L, Hammadi A, Hoyas-Sanchez C, Jimenez-Anton A, Almansa-Lopez A, Casares-Martin-Moreno L, Sanchez-Alvarez E, Murillo-Rodriguez A, Gomez-Mora M, Gomez-Pontes Cabrera T, Romero-Palacios PJ, Alcazar-Navarrete B. Short term exacerbation risk and exhaled nitric oxide in COPD. Respir Med. 2025 Jul;243:108134. doi: 10.1016/j.rmed.2025.108134. Epub 2025 Apr 30. PMID 40316031